CLINICAL TRIAL: NCT06715007
Title: Antiplatelet Therapy and Endothelial-stabilizing Agents in Cerebral Small Vessel Diseases
Acronym: Athena-cSVD
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Wang Zhaolu, Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: Athena-cSVD
Record Dates: First submitted 2023-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Small Vessel Cerebrovascular Disease; White Matter Hyperintensity
Keywords: cerebral small vessel disease; White Matter Hyperintensity; recent small subcortical infarcts; Endothelial dysfunction; cilostazol
MeSH Terms: conditions — Ischemic Stroke; Cerebral Small Vessel Diseases | interventions — Clopidogrel; Aspirin; Cilostazol; isosorbide-5-mononitrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with recent small subcortical infarct: Patient in this group will receive antiplatelet treatment (e.g. Aspirin, Clopidogrel, or Cilostazol),
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: Cilostazol + Isosorbide Mononitrate
- Patients with Whiter matter changes: White matter hyperintensities with a 2-3 grading on Fazekas scale will be recruited. Patient in this group will receive antiplatelet treatment (e.g. Aspirin, Clopidogrel, or Cilostazol),
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: Cilostazol + Isosorbide Mononitrate

INTERVENTIONS:
Drug: Clopidogrel — Patients will take Clopidogrel
Drug: Aspirin — Patients will take Rivaroxaban
Drug: Cilostazol + Isosorbide Mononitrate — Patients will take Cilostazol plus Isosorbide Mononitrate

SUMMARY:
Cerebral small vessel disease (cSVD) is a common accompaniment of aging. Recent small subcortical (or lacunar) infarcts (i.e. symptomatic cSVD) and white matter hyperintensities are typical cSVD lesions on neuroimaging. cSVD causes about a quarter of ischaemic strokes and related with cognitive dysfunction. However, few studies are available so far to especially explore the treatment of cSVD. Endothelial dysfunction plays an important part in cSVD. Cilostazol and isosorbide mononitrate have endothelial protective function. We designed this prospective cohort study in China, aiming to evaluate the effect of different antiplatelet agents (e.g. Cilostazol) on cSVD and retina in patients with cSVD (recent small subcortical infarcts or WMH, respectively).

DETAILED DESCRIPTION:
Cerebral small vessel disease (cSVD) is a common accompaniment of aging. It refers to a group of pathological processes with various etiologies that affect the small arteries, arterioles, venules, and capillaries of the brain. On neuroimaging, notably on magnetic resonance imaging (MRI), SVD has several visible signs, including recent small subcortical infarcts (i.e symptomatic cSVD in our study), lacunes of presumed vascular origin; white matter hyperintensities (WMH), perivascular spaces, cerebral microbleeds, cerebral microinfarcts and brain atrophy. SVD causes about a quarter of ischaemic strokes, is the main cause of vascular dementia, often occurs with Alzheimer's disease, contributing to about 50% of dementias worldwide. Although previous studies recommend BP control and antiplatelet therapy in symptomatic cSVD, secondary prevention strategies are mostly inferred from studies of ischemic stroke in general, the majority of which did not specifically investigate patients with symptomatic cSVD. In addition, long term dual antiplatelet therapy using clopidogrel and aspirin was shown to increase the risk of hemorrhage stroke in symptomatic cSVD, without any decrease in recurrent ischemic stroke.

Endothelial dysfunction plays an important part in cSVD. In addition to mild antiplatelet effects through the increase of cyclic adenosine monophosphate (cAMP), the phosphodiesterase (PDE) 3' inhibitor cilostazol is shown to be endothelial protective by several pathways, such as activation of endothelial nitric oxide (NO) synthase (NOS), regulation of endothelin-1. Isosorbide mononitrate (ISMN) is a NO donor, by augmenting the NO-cyclic guanosinemonophosphate phosphodiesterase-inhibitor pathway. Recent trial showed that the combined use of ISMN plus cilostazol was well tolerated and safe, and may reduce recurrent stroke and cognitive impairment after lacunar stroke.

Brain and retina possess numerous anatomical and functional similarities. Retinal capillary microvessels revealed by optical coherence tomography angiography (OCTA) have been found to be related to brain microvessels, reflecting the burden of cSVD. Retinal perfusion is also linked with cognitive function.

This cohort study will prospectively evaluate the effect of different antiplatelet agents on cSVD and retina in patients with cSVD (recent small subcortical infarcts or WMH, respectively).

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 30 years and ≤ 79 years.
2. A recent small subcortical infarct that occurred within 3 weeks prior to randomization; or patient with whiter matter hyperintensities with a 2-3 grading on Fazekas scale.
3. Absence of signs or symptoms of cortical dysfunction, such as aphasia, apraxia, agnosia, agraphia, homonymous visual field defect.
4. Modified Rankin score of ≤ 4.
5. In the absence of any other pathology in the parent artery at the site of the origin of the penetrating artery (focal atheroma, parent vessel dissection, vasculitis, vasospasm, and so on).

7. No ipsilateral cervical carotid stenosis (≥30%) by brain high resolution magnetic resonance imaging (HRMRI) or computed tomography angioplasty (CTA) or (magnetic resonance angioplasty) MRA and cervical artery ultrasound, if qualifying event is hemispheric. No vertebra artery stenosis (≥30%) by brain HRMRI or CTA or MRA and cervical artery ultrasound, if the lesion is in the territory of posterior circulation.

8. No major-risk cardioembolic sources requiring anticoagulation or other specific therapy.

9. Patient agrees with follow-up visits and is available by phone. 10. Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.

Exclusion criteria:

1. Intracranial aneurysms that need surgical treatment. Other significant active neurological illness e.g seizures, multiple sclerosis, intracranial tumor (except meningioma) or any intracranial vascular malformation.
2. Active cardiac disease (atrial fibrillation, myocardial infarct in last six months, active angina, symptomatic cardiac failure).
3. History of any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural).
4. Known allergy or contraindication to aspirin, clopidogrel, cilostazol, isosorbide mononitrate or statin.
5. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets < 100,000, hematocrit < 30, international normalized ratio (INR) > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), severe liver impairment (aspartate transaminase [AST] or alanine transaminase [ALT] > 3 x normal, cirrhosis), creatine kinase > 5 times the upper limit of normal (ULN) at final screening, severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) < 20mL/min/1.73 square meter at final screening.
6. Major surgery (including open femoral, aortic, cardiac or carotid surgery) within previous 30 days or planned in the 1 year after enrollment.
7. Dementia or psychiatric problem that prevents the patient from relevant evaluation or follow-up reliably.
8. Co-morbid conditions that may limit survival to less than 1 year.
9. Currently breastfeeding, pregnancy, planning to become pregnant and unwilling to use contraception for the duration of this study
10. Unable to tolerate, or contraindication to, MRI.
11. Enrollment in another study that would conflict with the current study.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a recent small subcortical infarct that occurred within 3 weeks prior to randomization， or patient with whiter matter hyperintensities with a 2-3 grading on Fazekas scale will be recruited.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
the impact of different antiplatelet agents on retinal vasculature. | 6 months follow up
  retinal vasculature will be assessed by optical coherence tomography and optical coherence tomography angiography.

SECONDARY OUTCOMES:
systemic or intracranial bleeding | systemic or intracranial bleeding will be assessed during 6 month follow-up.
occurrence of ischemic stroke or transient ischemic attack | during 6 month follow-up
Neurological function | Neurological function will be assessed at baseline, 1 week, 3 months and 6-month after recruitment.
  Neurological function will be assessed by NIHSS (National institute of health stroke scale)
Brain MRI (magnetic resonance imaging) | Brain MR will be performed at baseline and at 6 months after recruitment
  Brain MRI to evaluate whiter matter hyperintensities.
Cognitive function | MoCA will be assessed at baseline and at 3 and 6 months after recruitment.
  Montreal cognitive assessment (MoCA) will be used.
modified Rankin Scale (mRS) score | modified Rankin Scale (mRS) score will be assessed at baseline and at 3 and 6 months after recruitment.
Barthel index for activities of daily living | Barthel index will be assessed at baseline, 3 and 6 months after recruitment.
  Barthel index for activities of daily living is an ordinal scale which measures a person's ablility to complete activities of of daily living.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | UPDRS score will be evaluated at baseline and 3, 6 months after recruitment.
  MDS-UPDRS is scale to evaluate various aspects Parkinson's disease or Parkinsonism including non-motor and motor experiences of daily living and motor complications. Small vessel diseases may cause Parkinsonism, we thus use this scale in our study.

CONTACTS AND LOCATIONS:
Overall Officials: zhaolu wang, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China